CLINICAL TRIAL: NCT06489704
Title: Comparative Study of Pulmonary Artery Pressure (PAP) Assessed by Echocardiography in Patients With High Altitude Pulmonary Hypertension (HAPH) Permanently Residing Above 2500 Meters When Assessed Near Resident High Altitude (HA) at 3200 m vs. at Low Altitude (LA) at 760 m
Brief Title: High Altitude (HA) Residents With High Altitude Pulmonary Hypertension (HAPH), Pulmonary Artery Pressure (PAP) Assessed at HA (3200 m) vs LA (760 m)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HAPH_HAvsLA_PAP
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; High Altitude; Pulmonal Arterial Pressure
MeSH Terms: conditions — Pulmonary edema of mountaineers; Hypertension, Pulmonary; Hypoxia; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Each highlander with HAPH will perform a echocardiography at high altitude (HA, 3200 m) and day 2 and day 7 at low altitude (LA, 760 m) according to a prospective study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessments at 3200 m and 760 m, respectively (Experimental): Participants will have a echocardiography near their resident altitude at 3200 m and after relocation to 760 m after 1 and 7 days
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Echocardiography will be performed according to clinical standards

SUMMARY:
To study the effect of relocation from 3200 m (Aksay) to 760 m (Bishkek) in patients with high altitude pulmonary hypertension (HAPH) who permanently live >2500 m on pulmonary artery pressure (PAP)

DETAILED DESCRIPTION:
This research in highlanders with HAPH diagnosed by echocardiography and defined by a RV/RA >30 mmHg who permanently live at HA >2500 m will have pulmonary arterial pressure (PAP) assessed by echocardiography near their living altitude in Aksay at 3200 m and at 760 m in Bishkek the day after the first and the seventh night after relocation.

ELIGIBILITY:
Inclusion Criteria:

* Permanently living >2500 m
* HAPH diagnosed with a minimum RV/RA of 30 mmHg assessed by echocardiography at an altitude of 3200 m
* Written informed consent

Exclusion Criteria:

* Highlanders who cannot follow the study investigations,
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, heavy smoking >20 cigarettes/day or >20 pack-years.
* Coexistent unstable systemic hypertension or coronary artery disease that required adjustment of medication within the last 2 months
* Regular use of medication that affects control of breathing (benzodiazepines, opioids, acetazolamide)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary artery Pressure (PAP) after the first night at 760 m (LA) vs at 3200 m (HA) | day 2 at 760 m vs. 3200 m
  Change in RV/RA in mmHg assessed by echocardiography between LA (760 m) vs High altitude (3200 m)

SECONDARY OUTCOMES:
Change in Pulmonary artery Pressure (PAP) after seven nights at 760 m (LA) vs at 3200 m (HA) | day 7 at 760 m vs. 3200 m
  Change in RV/RA in mmHg assessed by echocardiography between LA (760 m) vs High altitude (3200 m)
Cardiac output at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Change in cardiac output in l/min assessed by echocardiography between LA (760 m) vs HA (3200 m)
Tricuspid pressure gradient by echocardiography at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Tricuspid pressure gradient assessed by echocardiography between LA (760 m) vs HA (3200 m)
Tricupsid annular plane systolic excursion by echocardiography at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Tricupsid annular plane systolic excursion assessed by echocardiography between LA (760 m) vs HA (3200 m)
pH by arterial blood gases at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Change in pH by arterial blood gases assessed between LA (760 m) vs HA (3200 m)
partial pressure of oxygen (PaO2) by arterial blood gases at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Change in partial pressure of oxygen (PaO2) assessed by arterial blood gases between LA (760 m) vs HA (3200 m)
partial pressure of carbon dioxide (PaCO2) by arterial blood gases at 760 m (LA) vs at 3200 m (HA) | after the first and seventh night at LA
  Change in partial pressure of carbon dioxide (PaCO2) assessed by arterial blood gases partial pressure of carbon dioxide (PaCO2) between LA (760 m) vs HA (3200 m)
Change in right to left heart diameter ratio at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Change in right to left heart diameter ratio assessed by echocardiography between LA (760 m) vs HA (3200 m)
Change in right atrial area at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Change in right atrial area by echocardiography between LA (760 m) vs HA (3200 m)
Change in right heart strain at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Change in right heart strain by echocardiography between LA (760 m) vs HA (3200 m)
Change in ECG morphology at 760 m (LA) vs at 3200 m (HA) | day 2 and 7 at 760 m vs. 3200 m
  Change in ECG morphology and QT-interval by 12-lead ECG between LA (760 m) vs HA (3200 m)

CONTACTS AND LOCATIONS:
Overall Officials: Talant M Sooronbaev, Prof. Dr., Principal Investigator — National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov; Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- Aksay Medical Center, Aksay Plateau, Naryn, Kyrgyzstan, Kyrgyzstan, Kyrgyzstan